CLINICAL TRIAL: NCT01721616
Title: A Randomized Clinical Trial of Cefazolin Versus Cefazolin Plus Azithromycin Prophylaxis in Post-Cesarean Endometritis
Brief Title: Comparison Study of Cefazolin Versus Cefazolin Plus Azithromycin Prophylaxis in Post-Cesarean Endometritis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Pedro Morales-Ramirez, MD, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 12-13
Record Dates: First submitted 2012-11-01; First posted 2012-11-06 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Endometritis
MeSH Terms: conditions — Endometritis | interventions — Azithromycin; Cefazolin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cefazolin (Active Comparator): single antibiotic
  Interventions: Drug: Cefazolin
- Cefazolin + Azitrhromycin (Active Comparator): double antibiotic
  Interventions: Drug: Azithromycin; Drug: Cefazolin

INTERVENTIONS:
Drug: Azithromycin
  Arms: Cefazolin + Azitrhromycin
Drug: Cefazolin

SUMMARY:
Despite the generalized use of preoperative antibiotic prophylaxis, endometritis remains as the most frequent post-cesarean delivery complication. This increased morbidity translates into extended post-partum antibiotic use and prolongation of hospital stay with the subsequent increase in health care expenses. The current regimen recommended by the American College of Obstetricians and Gynecologists for cesarean delivery prophylaxis (1st generation cephalosporins) does not cover for Ureaplasma Urealyticum, a microorganism that has been associated with an increased risk of endometritis in post-cesarean section patients. Azithromycin, an antibiotic that has both aerobic and some anaerobic coverage, uniquely covers Ureaplasma and would be an excellent second antibiotic for cesarean section chemoprophylaxis. Our hypothesis is that the addition of azithromycin to standard chemoprophylaxis with cefazolin can effect a 25% reduction of post-cesarean section endometritis.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients between 37 and 42 weeks gestational weeks.
* Pregnant patients undergoing indicated cesarean section at Truman Medical Center Hospital July 2012 and July 2014.
* Pregnant patient that received prenatal care at Truman Medical Center. Hospital Hill, Samuel Rogers or Swope Parkway health centers at least 1 month prior to the Cesarean delivery.
* Signed informed consent.

Exclusion Criteria:

* Allergy to cephalosporins or azithromycin.
* Refusal to sign consent form.
* Clinical signs of chorioamnionitis: fever 100.4 F or higher, uterine tenderness, maternal or fetal tachycardia.
* Immunocompromised condition: HIV positive with CD4 count below 200, chronic steroid use, pregestational diabetes, cancer, chemotherapy.
* Need for emergent cesarean precluding consent or availability of study medication.
* Need for hysterectomy at cesarean section.
* Use of antibiotic in the 72 hours prior to admission.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Development of post cesarean endometritis | 3-4 days while in hospital during post partum period

SECONDARY OUTCOMES:
Hospital stay length | 3-4 days while in hospital during post partum period

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Morales, MD, Principal Investigator — University of Missouri, Kansas City; Katherine Goodpasture, DO, Principal Investigator — University of Missouri, Kansas City
Locations (1):
- Truman Medical Center - Hospital Hill, Kansas City, Missouri, United States